CLINICAL TRIAL: NCT02752997
Title: Reducing 30-day Readmissions in Patients With Heart Failure Through Pharmacist Discharge Medication Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sarah Lessard, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Factorial | Masking: None
Other Study IDs: 15-008286
Record Dates: First submitted 2016-04-14; First posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Heart Failure; Patient Readmission
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Discharge medication services included:
  * Discharge medication reconciliation
  * Identification of medication discrepancies and resolution
  * Medication counseling using health coaching techniques with short term goal setting and follow up phone call
  Interventions: Other: Pharmacist discharge medication services
- Comparator (No Intervention): Current standard of care provided by nursing staff.

INTERVENTIONS:
Other: Pharmacist discharge medication services — Included in arm descriptions
  Arms: Intervention

SUMMARY:
Patients admitted for heart failure that are provided discharge medication services by a pharmacist are less likely to be readmitted within 30 days of primary admission.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of heart failure, discharged from any medical service

Exclusion Criteria:

* Unwilling to participate, discharged to nursing/rehab facility, non-English speaking, resident unavailable

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of patients readmitted to the hospital within 30 days of primary heart failure admission | 30 Days
  Fisher's T-test

SECONDARY OUTCOMES:
Number of patients who visit the emergency department within 30 days of primary heart failure admission | 30 Days
  Fisher's T-test
Number of medication discrepancies identified and the number of medication discrepancies resolved by the pharmacist at discharge. | 30 Days
  Fisher's T-test
Number of short term goals set by patient's at discharge and the number of short term goals met by patient's at the 7-10 follow up phone call. | 30 days
  Number of short term goals set will be compared to the number of goals patients achieved, comparison will be calculated by percentage

CONTACTS AND LOCATIONS:
Overall Officials: Sarah R Lessard, Pharm.D., Principal Investigator — Mayo Clinic Health System - Franciscan Healthcare
Locations (1):
- Mayo Clinic Health System - Franciscan Healthcare, La Crosse, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bishop MA, Cohen BA, Billings LK, Thomas EV. Reducing errors through discharge medication reconciliation by pharmacy services. Am J Health Syst Pharm. 2015 Sep 1;72(17 Suppl 2):S120-6. doi: 10.2146/sp150021. PMID 26272892
- [Background] Dharmarajan K, Hsieh AF, Lin Z, Bueno H, Ross JS, Horwitz LI, Barreto-Filho JA, Kim N, Bernheim SM, Suter LG, Drye EE, Krumholz HM. Diagnoses and timing of 30-day readmissions after hospitalization for heart failure, acute myocardial infarction, or pneumonia. JAMA. 2013 Jan 23;309(4):355-63. doi: 10.1001/jama.2012.216476. PMID 23340637
- [Background] Dudas V, Bookwalter T, Kerr KM, Pantilat SZ. The impact of follow-up telephone calls to patients after hospitalization. Dis Mon. 2002 Apr;48(4):239-48. doi: 10.1016/s0011-5029(02)90031-3. PMID 12021756
- [Background] Emmons KM, Rollnick S. Motivational interviewing in health care settings. Opportunities and limitations. Am J Prev Med. 2001 Jan;20(1):68-74. doi: 10.1016/s0749-3797(00)00254-3. PMID 11137778
- [Background] Eggink RN, Lenderink AW, Widdershoven JW, van den Bemt PM. The effect of a clinical pharmacist discharge service on medication discrepancies in patients with heart failure. Pharm World Sci. 2010 Dec;32(6):759-66. doi: 10.1007/s11096-010-9433-6. Epub 2010 Sep 1. PMID 20809276
- [Background] Farris KB, Carter BL, Xu Y, Dawson JD, Shelsky C, Weetman DB, Kaboli PJ, James PA, Christensen AJ, Brooks JM. Effect of a care transition intervention by pharmacists: an RCT. BMC Health Serv Res. 2014 Sep 18;14:406. doi: 10.1186/1472-6963-14-406. PMID 25234932
- [Background] Gianos E, Schoenthaler A, Mushailov M, Fisher EA, Berger JS. Rationale and design of the Investigation of Motivational Interviewing and Prevention Consults to Achieve Cardiovascular Targets (IMPACT) trial. Am Heart J. 2015 Sep;170(3):430-7.e9. doi: 10.1016/j.ahj.2015.06.001. Epub 2015 Jun 6. PMID 26385025
- [Background] Gunadi S, Upfield S, Pham ND, Yea J, Schmiedeberg MB, Stahmer GD. Development of a collaborative transitions-of-care program for heart failure patients. Am J Health Syst Pharm. 2015 Jul 1;72(13):1147-52. doi: 10.2146/ajhp140563. PMID 26092965
- [Background] Hall MJ, Levant S, DeFrances CJ. Hospitalization for congestive heart failure: United States, 2000-2010. NCHS Data Brief. 2012 Oct;(108):1-8. PMID 23102190
- [Background] Harrison PL, Hara PA, Pope JE, Young MC, Rula EY. The impact of postdischarge telephonic follow-up on hospital readmissions. Popul Health Manag. 2011 Feb;14(1):27-32. doi: 10.1089/pop.2009.0076. Epub 2010 Nov 19. PMID 21090991
- [Background] Linden A, Butterworth SW, Prochaska JO. Motivational interviewing-based health coaching as a chronic care intervention. J Eval Clin Pract. 2010 Feb;16(1):166-74. doi: 10.1111/j.1365-2753.2009.01300.x. PMID 20367828
- [Background] May CS, Russell CS. Health coaching: adding value in healthcare reform. Glob Adv Health Med. 2013 May;2(3):92-4. doi: 10.7453/gahmj.2013.032. PMID 24416677
- [Background] Ni H, Xu J. Recent Trends in Heart Failure-related Mortality: United States, 2000-2014. NCHS Data Brief. 2015 Dec;(231):1-8. PMID 26727546
- [Background] Roger VL. Epidemiology of heart failure. Circ Res. 2013 Aug 30;113(6):646-59. doi: 10.1161/CIRCRESAHA.113.300268. PMID 23989710
- [Background] WRITING COMMITTEE MEMBERS; Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on practice guidelines. Circulation. 2013 Oct 15;128(16):e240-327. doi: 10.1161/CIR.0b013e31829e8776. Epub 2013 Jun 5. No abstract available. PMID 23741058
- [Background] Warden BA, Freels JP, Furuno JP, Mackay J. Pharmacy-managed program for providing education and discharge instructions for patients with heart failure. Am J Health Syst Pharm. 2014 Jan 15;71(2):134-9. doi: 10.2146/ajhp130103. PMID 24375606
- [Background] Szkiladz A, Carey K, Ackerbauer K, Heelon M, Friderici J, Kopcza K. Impact of pharmacy student and resident-led discharge counseling on heart failure patients. J Pharm Pract. 2013 Dec;26(6):574-9. doi: 10.1177/0897190013491768. PMID 23797199
- [Background] Stawnychy M, Masterson Creber R, Riegel B. Using brief motivational interviewing to address the complex needs of a challenging patient with heart failure. J Cardiovasc Nurs. 2014 Sep-Oct;29(5):E1-6. doi: 10.1097/JCN.0000000000000098. PMID 24231890
- [Background] Sarangarm P, London MS, Snowden SS, Dilworth TJ, Koselke LR, Sanchez CO, D'Angio R, Ray G. Impact of pharmacist discharge medication therapy counseling and disease state education: Pharmacist Assisting at Routine Medical Discharge (project PhARMD). Am J Med Qual. 2013 Jul-Aug;28(4):292-300. doi: 10.1177/1062860612461169. Epub 2012 Oct 2. PMID 23033542
- [Background] Salvo MC, Cannon-Breland ML. Motivational interviewing for medication adherence. J Am Pharm Assoc (2003). 2015 Jul-Aug;55(4):e354-61; quiz e362-3. doi: 10.1331/JAPhA.2015.15532. PMID 26161493
- [Background] Salas CM, Miyares MA. Implementing a pharmacy resident run transition of care service for heart failure patients: Effect on readmission rates. Am J Health Syst Pharm. 2015 Jun 1;72(11 Suppl 1):S43-7. doi: 10.2146/sp150012. PMID 25991595
- [Background] Wang H, Robinson RD, Johnson C, Zenarosa NR, Jayswal RD, Keithley J, Delaney KA. Using the LACE index to predict hospital readmissions in congestive heart failure patients. BMC Cardiovasc Disord. 2014 Aug 7;14:97. doi: 10.1186/1471-2261-14-97. PMID 25099997
- [Background] Albert NM, Barnason S, Deswal A, Hernandez A, Kociol R, Lee E, Paul S, Ryan CJ, White-Williams C; American Heart Association Complex Cardiovascular Patient and Family Care Committee of the Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Quality of Care and Outcomes Research. Transitions of care in heart failure: a scientific statement from the American Heart Association. Circ Heart Fail. 2015 Mar;8(2):384-409. doi: 10.1161/HHF.0000000000000006. Epub 2015 Jan 20. PMID 25604605
- See also: Centers for Medicare and Medicaid Services Website — https://www.cms.gov/medicare/medicare-fee-for-service-payment/acuteinpatientpps/readmissions-reduction-program.html
- See also: Centers for Medicare and Medicaid Services Website — https://www.cms.gov/Medicare/Medicare-Fee-for-Service-Payment/AcuteInpatientPPS/index.html